CLINICAL TRIAL: NCT02748889
Title: An Open Label, Randomized Phase I/II Trial of Carboplatin Plus Etoposide With ot Without MPDL3280A in Untreated Extensive Stage Small Cell Lung Cancer
Brief Title: Carboplatin Plus Etoposide With or Without MPDL3280A in Untreated Extensive Stage Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Difficulties with recruitment
Sponsor: Giuseppe Giaccone (Other)
Collaborators: Vanderbilt University (Other); Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor-Investigator, Giuseppe Giaccone, Associate Director for Clinical Research, Georgetown University
Organization: Georgetown University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-1380
Record Dates: First submitted 2016-02-02; First posted 2016-04-22 (Estimated); Results first posted 2018-07-02 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Small Cell Lung Cancer ( SCLC )
Keywords: SCLC; Small Cell; Lung Cancer; MPDL3280A; atezolizumab
MeSH Terms: conditions — Small Cell Lung Carcinoma; Lung Neoplasms | interventions — Carboplatin; Etoposide; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Carboplatin plus etoposide (Active Comparator): Carboplatin AUC 5 iv on day 1 every 21 days for 4 cycles Etoposide 100mg/m2 iv on days 1-3 every 21 days for 4 cycles
  Interventions: Drug: Carboplatin; Drug: Etoposide
- Carboplatin, etoposide and MPDL3280A (Experimental): Carboplatin AUC 5 iv on day 1 every 21 days for 4 cycles Etoposide 100mg/m2 iv on days 1-3 every 21 days for 4 cycles MPDL3280A (Atezolizumab) 1200mg iv on day 1 every 21 days until progression
  Interventions: Drug: Carboplatin; Drug: Etoposide; Biological: MPDL3280A

INTERVENTIONS:
Drug: Carboplatin — Standard chemotherapy
  Other Names: Paraplatin
Drug: Etoposide — Standard chemotherapy
  Other Names: VP-16, Toposar
Biological: MPDL3280A — Experimental biologic
  Other Names: Atezolizumab
  Arms: Carboplatin, etoposide and MPDL3280A

SUMMARY:
This is an open-label study with two parts, a Phase I study and a randomized Phase II study. This study will be conducted at approximately ten sites in the United States. Approximately 178 patients will be enrolled in this trial.

DETAILED DESCRIPTION:
Combining standard chemotherapy with a PD-1/PD-L1 inhibitor holds great appeal in the treatment of SCLC. While this approach may be appropriate for many cancer types, SCLC may be particularly vulnerable to this treatment strategy. Early studies have suggested greater efficacy with agents targeting PD-1/PD-L1 in tumors that are more mutationally complex, such as those associated with tobacco use. SCLC has a strong association with tobacco use and indeed, genome-wide sequencing studies have consistently shown that SCLC carries one of the highest rates of non-synonymous mutations. In addition, MPDL3280A has been safely combined with platinum based chemotherapy doublets in the treatment of NSCLC. Thus, a combination of carboplatin, etoposide and MPDL3280A may significantly improve outcomes in the treatment of SCLC.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form (ICF)
* Ability and willingness to comply with the requirements of the study protocol
* Age 18 years or older
* Histological or cytological diagnosis of ES-SCLC (Note: Extensive-stage disease is defined as disease beyond the ipsilateral hemithorax, mediastinum and ipsilateral supraclavicular area and including malignant pleural or pericardial effusion or hematogenous metastases)
* Patients with mixed histology SCLC and NSCLC are permitted
* Representative tumor specimens in paraffin blocks (preferred) or at least 10 unstained slides, with an associated pathology report, requested at any time prior to study entry. Tissue from core needle, punch, or excisional biopsy sample collection is preferred but slides from fine needle aspiration, brushing, and lavage samples are acceptable.
* Adequate hematologic and end organ function, defined by the following laboratory results obtained within 14 days prior to the first study treatment (Cycle 1, Day 1)
* ANC 1000 cells/mL
* WBC counts 2500/mL
* Lymphocyte count 500/mL
* Platelet count 100,000/mL
* Hemoglobin 9.0 g/dL (transfusion to meet this criterion is permitted)
* Serum sodium greater than 120 mmol/L
* Total bilirubin must be 1.5 ULN with the following exception:

Patients with known Gilbert disease who have serum bilirubin level 3 ULN may be enrolled.

- AST and ALT 3.0 ULN with the following exception: Patients with liver involvement: AST and/or ALT 5 ULN

- Alkaline phosphatase 2.5 ULN with the following exception:

Patients with liver or bone inv ULN or creatinine clearance 50 mL/min on the basis of the Cockcroft-Gault glomerular filtration rate estimation:

(140 age) (weight in kg) (0.85 if female) 72 (serum creatinine in mg/dL)

* Measurable disease per RECIST v1.1 (see Appendix 6)
* Patients with asymptomatic CNS metastases are allowed
* For female patients of childbearing potential and male patients with partners of childbearing potential, agreement (by patient and/or partner) to use highly effective form(s) of contraception (i.e., one that results in a low failure rate [ 1 percent per year] when used consistently and correctly) and to continue its use for 6 months after the last dose of MPDL3280A
* ECOG performance status of 0 or 1 (see Appendix 8)
* Patients with ECOG performance status of 2, secondary to the underlying disease, may be enrolled in the Phase II portion of the study
* INR and aPTT within 1.5 ULN
* This applies only to patients who do not receive therapeutic anticoagulation; patients receiving therapeutic anticoagulation (such as low molecular weight heparin or warfarin) should be on a stable dose.

Exclusion Criteria:

* Inability to comply with study and follow-up procedures
* Limited stage SCLC appropriate for definitive treatment with chemoradiation
* Prior systemic anti-cancer therapy for small cell lung cancer
* Prior palliative radiation therapy less than 2 weeks prior to administration of study treatment or prior whole brain radiation therapy (WBRT) less than 4 weeks prior to study treatment
* Symptomatic brain metastases (patients with asymptomatic brain metastases may be eligible provided other criteria are met)
* Leptomeningeal disease or carcinomatous meningitis
* Uncontrolled hypercalcemia ( ≥1.5 mmol/L ionized calcium or Ca > 12 mg/dL) or symptomatic hypercalcemia requiring continued use of bisphosphonate therapy or denosumab (patients receiving bisphosphonate therapy or denosumab to prevent skeletal events and who do not have a history of clinically significant hypercalcemia are eligible, though patients receiving denosumab must be willing and eligible to receive bisphosphonates instead)
* Malignancies other than SCLC within 2 years prior to administration of study treatment with the exception of those with a negligible risk of metastases or death treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix or breast, basal or squamous cell skin cancer, or localized prostate cancer treated definitively)
* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis, cirrhosis, fatty liver, and inherited liver disease
* Pregnancy, lactation, or breastfeeding
* History or risk of autoimmune disease, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjogren's syndrome, Bell's palsy, Guillain-Barré syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, or glomerulonephritis
* Patients with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone may be eligible.
* Patients with controlled Type 1 diabetes mellitus on a stable insulin regimen may be eligible.
* Patients with eczema, psoriasis, lichen simplex chronicus of vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions:
* Patients with psoriasis must have a baseline ophthalmologic exam to rule out ocular manifestations
* Rash must cover less than 10% of body surface area (BSA)
* Disease is well controlled at baseline and only requiring low potency topical steroids (e.g., hydrocortisone 2.5%, hydrocortisone butyrate 0.1%, flucinolone 0.01%, desonide 0.05%, aclometasone dipropionate 0.05%)
* No acute exacerbations of underlying condition in the last 12 months (not requiring PUVA [psoralen plus ultraviolet A radiation], methotrexate, retinoids, biologics, oral calcineurin inhibitors, high potency oral steroids)
* History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest CT scan
* History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* History of HIV infection or active hepatitis B (chronic or acute) or hepatitis C infection
* Patients with past or resolved hepatitis B infection (defined as having a negative hepatitis B surface antigen [HBsAg] test and a positive anti-HBc [antibody to hepatitis B core antigen] antibody test) are eligible.
* Patients positive for HCV antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
* Active, clinically serious infections of NCI CTCAE v4.0 Grade 2 or higher within 4 weeks prior to Cycle 1, Day 1
* Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction within the previous 3 months, unstable arrhythmias, or unstable angina. Patient with known coronary artery disease, congestive heart failure not meeting the above criteria, or known left ventricular ejection fraction less than 50% must be on a stable medical regimen that is optimized in the opinion of the treating physician
* Major surgical procedure within 28 days prior to Cycle 1, Day 1 or anticipation of need for a major surgical procedure during the course of the study
* History of stroke or transient ischemic attack (TIA) within 6 months prior to Cycle 1, Day 1
* Administration of a live, attenuated vaccine within 4 weeks before Cycle 1, Day 1 or anticipation that such a live attenuated vaccine will be required during the study
* Influenza vaccination should be given during influenza season only (approximately October to March). Patients must not receive live, attenuated influenza vaccine (e.g., FluMist) within 4 weeks prior to Cycle 1, Day 1 or at any time during the study.
* Treatment with systemic immunostimulatory agents (including but not limited to IFN , IL-2) within 6 weeks or five half-lives of the drug (whichever is shorter) prior to Cycle 1, Day 1
* Prior treatment with antiPD-1, or antiPD-L1 therapeutic antibody or pathway targeting agents
* Patients who have received prior treatment with antiCTLA-4 may be enrolled, provided the following requirements are met:
* Minimum of 12 weeks from the first dose of antiCTLA-4 and 6 weeks from the last dose
* No history of severe immune-related adverse effects from anti CTLA 4 (CTCAE Grade 3 and 4)
* Treatment with investigational agent within 4 weeks prior to Cycle 1, Day 1 (or within five half lives of the investigational product, whichever is longer)
* Treatment with systemic immunosuppressive medications (including but not limited to prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti tumor necrosis factor [TNF] agents) within 2 weeks prior to Cycle 1, Day 1
* Patients who have received acute, low dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled.
* The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed.
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* Patients with prior allogeneic bone marrow transplantation or prior solid organ transplantation
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-05-09 (Actual); Study Completion 2017-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe ( Beppe) Giaccone, Md,PhD, Study Chair — Georgetown Lombardi Comprehensive Cancer Center
Locations (1):
- Georgetown Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rossi A, Di Maio M, Chiodini P, Rudd RM, Okamoto H, Skarlos DV, Fruh M, Qian W, Tamura T, Samantas E, Shibata T, Perrone F, Gallo C, Gridelli C, Martelli O, Lee SM. Carboplatin- or cisplatin-based chemotherapy in first-line treatment of small-cell lung cancer: the COCIS meta-analysis of individual patient data. J Clin Oncol. 2012 May 10;30(14):1692-8. doi: 10.1200/JCO.2011.40.4905. Epub 2012 Apr 2. PMID 22473169
- [Background] Blank C, Gajewski TF, Mackensen A. Interaction of PD-L1 on tumor cells with PD-1 on tumor-specific T cells as a mechanism of immune evasion: implications for tumor immunotherapy. Cancer Immunol Immunother. 2005 Apr;54(4):307-14. doi: 10.1007/s00262-004-0593-x. Epub 2004 Dec 15. PMID 15599732
- [Background] Blank C, Mackensen A. Contribution of the PD-L1/PD-1 pathway to T-cell exhaustion: an update on implications for chronic infections and tumor evasion. Cancer Immunol Immunother. 2007 May;56(5):739-45. doi: 10.1007/s00262-006-0272-1. Epub 2006 Dec 29. PMID 17195077
- [Background] Brahmer J, Reckamp KL, Baas P, Crino L, Eberhardt WE, Poddubskaya E, Antonia S, Pluzanski A, Vokes EE, Holgado E, Waterhouse D, Ready N, Gainor J, Aren Frontera O, Havel L, Steins M, Garassino MC, Aerts JG, Domine M, Paz-Ares L, Reck M, Baudelet C, Harbison CT, Lestini B, Spigel DR. Nivolumab versus Docetaxel in Advanced Squamous-Cell Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Jul 9;373(2):123-35. doi: 10.1056/NEJMoa1504627. Epub 2015 May 31. PMID 26028407
- [Background] Segal, N.H., et al., Preliminary data from a multi-arm expansion study of MEDI4736, an anti-PD-L1 antibody. J Clin Oncol, 2014. 32(5S): p. abstr 3002
- [Background] Lutzky, J., et al., A phase 1 study of MEDI4736, an anti-PD-L1 antibody, in patients with advanced solid tumors. J Clin Oncol, 2014. 32(5S): p. abstr 3001
- [Background] Antonia, S.J., et al., Phase I/II study of nivolumab with or without ipilimumab for treatment of recurrent small cell lung cancer (SCLC): CA209-032. J Clin Oncol, 2015. 33: p. abstr 7503
- [Background] Brahmer JR, Tykodi SS, Chow LQ, Hwu WJ, Topalian SL, Hwu P, Drake CG, Camacho LH, Kauh J, Odunsi K, Pitot HC, Hamid O, Bhatia S, Martins R, Eaton K, Chen S, Salay TM, Alaparthy S, Grosso JF, Korman AJ, Parker SM, Agrawal S, Goldberg SM, Pardoll DM, Gupta A, Wigginton JM. Safety and activity of anti-PD-L1 antibody in patients with advanced cancer. N Engl J Med. 2012 Jun 28;366(26):2455-65. doi: 10.1056/NEJMoa1200694. Epub 2012 Jun 2. PMID 22658128
- [Background] Reck M, Bondarenko I, Luft A, Serwatowski P, Barlesi F, Chacko R, Sebastian M, Lu H, Cuillerot JM, Lynch TJ. Ipilimumab in combination with paclitaxel and carboplatin as first-line therapy in extensive-disease-small-cell lung cancer: results from a randomized, double-blind, multicenter phase 2 trial. Ann Oncol. 2013 Jan;24(1):75-83. doi: 10.1093/annonc/mds213. Epub 2012 Aug 2. PMID 22858559
- [Background] Liu, S.V., et al., Safety and efficacy of MPDL3280A (anti-PDL1) in combination with platinum-based doublet chemotherapy in patients with advanced non-small cell lung cancer (NSCLC). J Clin Oncol, 2015. 33: p. abstr 8030
- [Background] Powderly, J.D., et al., Biomarkers and associations with the clinical activity of PD-L1 blockade in a MPDL3280A study. J Clin Oncol, 2013. suppl; abstr 3001

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Carboplatin Plus Etoposide | Carboplatin, Etoposide and MPDL3280A
Started | 0 | 1
Completed | 0 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This study enrolled one subject before being terminated early due to recruitment difficulties.That subject was assigned to the Carboplatin, Etoposide, and MPDL3280A arm. No subjects were enrolled to the Carboplatin and Etoposide arm
Groups:
- Total: Total of all reporting groups
Arm/Group | Carboplatin Plus Etoposide | Carboplatin, Etoposide and MPDL3280A | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 0 | 0
  Between 18 and 65 years |  | 1 | 1
  >=65 years |  | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] |  | 58 (0) | 58 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 0 | 0
  Male |  | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0
  Asian |  | 0 | 0
  Native Hawaiian or Other Pacific Islander |  | 0 | 0
  Black or African American |  | 1 | 1
  White |  | 0 | 0
  More than one race |  | 0 | 0
  Unknown or Not Reported |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) With Carboplatin, Etoposide and MPDL3280A Compared to Chemotherapy Alone According to RECIST v1.1
Description: Disease progression will be assessed per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT and bone scans.
Time Frame: From the first occurrence of progression or death, whichever occurred first, assessed up to 2 years.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Carboplatin, Etoposide and MPDL3280A
Number analyzed (Participants) | 1
months | 6 (0)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for each subject from the time they signed the informed consent until study completion. The period of collection depended on the length of the treatment period. For the single subject enrolled, this amounted to 6.5 months.
Arm/Group | Carboplatin, Etoposide and MPDL3280A
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carboplatin, Etoposide and MPDL3280A (N=1)
Headache (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carboplatin, Etoposide and MPDL3280A (N=1)
Infusion reaction (General disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 1 (1)
Headache (General disorders) | 1 (1)
Myalgias (Musculoskeletal and connective tissue disorders) | 1 (1)
Night Sweats (General disorders) | 1 (1)
Hypophosphatemia (Blood and lymphatic system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Hypoalbuminemia (Hepatobiliary disorders) | 1 (1)
Hypokalemia (Blood and lymphatic system disorders) | 1 (1)
Increased bilirubin (Hepatobiliary disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Neuropathy (Nervous system disorders) | 1 (1)
ALT Elevation (Hepatobiliary disorders) | 1 (1)
Dizziness (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-13): https://cdn.clinicaltrials.gov/large-docs/89/NCT02748889/Prot_SAP_000.pdf